CLINICAL TRIAL: NCT01634542
Title: A Non-Interventional Prospective Cohort Study of Patients With Persistent Symptoms of Schizophrenia to Describe The Course and Burden of Illness
Brief Title: An Non-Interventional Study of Patients With Persistent Symptoms of Schizophrenia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MN28151
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, prospective, non-interventional study will evaluate the prevalence and characteristics of patients with persistent symptoms of schizophrenia and the course of their illness over 24 months.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adult patients, >/= 18 years of age
* Diagnosis of schizophrenia according to Diagnostic and Statistical Manual for Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) or International Classification of Diseases, 10th revision (ICD-10)

Caregivers:

* Age >/= 18 years
* Family member or friend of the patient, who spends at least 4 hours a week with the patient

Exclusion Criteria:

* Acute psychotic exacerbation in the 3 months prior to the baseline observation (e.g. hospitalization or increased psychiatric care in order to prevent hospitalization)
* Enrolled in an interventional study at the baseline observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent symptoms of schizophrenia
Sampling Method: Probability Sample
Enrollment: 1433 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Course of illness: Change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scores | from baseline to Month 24

SECONDARY OUTCOMES:
Frequency/characteristics (PANSS) of patients with diagnosis of schizophrenia of >/= 12 months duration before baseline | at screening (approximately 18 months)
Duration/severity of symptoms of schizophrenia according to Personal Social Performance Scale (PSP) / Health Related Quality of Life (HRQoL) questionnaire | 24 months
Medical resource utilization/costs | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (125):
- Argentina (3):
  - Buenos Aires
  - Caba
  - La Plata
- Brazil (3):
  - Goiânia, Goiás
  - Curitiba, Paraná
  - São Paulo, São Paulo
- Canada (8):
  - Medicine Hat, Alberta
  - Vancouver, British Columbia
  - Chatam, Ontario
  - Mississauga, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Verdun, Quebec
- France (21):
  - Aix-en-Provence
  - Chaumont
  - Colmar
  - Corbeil-Essonnes
  - Issy-les-Moulineaux
  - Lille
  - Lyon
  - Marseille
  - Montberon
  - Montebeliard
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Poitiers
  - Rennes
  - Rouffach
  - Saint-Cyr-au-Mont-d'Or
  - Tassin-la-Demi-Lune
  - Toulouse
  - Verdun
- Germany (30):
  - Aachen
  - Alzey
  - Augsburg
  - Bad Zwischenahn
  - Berlin
  - Bochum
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Ellwangen
  - Essen
  - Grünstadt
  - Halle
  - Hamburg
  - Homburg/Saar
  - Jena
  - Koeln-Pulheim
  - Leipzig
  - Magdeburg
  - Mainz
  - Mannheim
  - Marburg
  - Mittweida
  - Oranienburg
  - Regensburg
  - Rostock
  - Siegen
  - Weinsberg
  - Westerstede
- Italy (22):
  - Bari, Apulia
  - Catanzaro, Calabria
  - Bologna, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Cassina Nuova Di Bollate, Lombardy
  - Gardone V.T., Lombardy
  - Milan, Lombardy
  - Campobasso, Molise
  - Bra, Piedmont
  - Novara, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Florence, Tuscany
  - Perugia, Umbria
  - Conegliano, Veneto
  - Padua, Veneto
- Spain (23):
  - Alcoy, Alicante
  - Almería, Almeria
  - Manacor, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Burgos, Burgos
  - Santander, Cantabria
  - Torrelavega, Cantabria
  - Granada, Granada
  - A Coruña, La Coruña
  - Málaga, Malaga
  - Pamploma, Navarre
  - Pamplona, Navarre
  - Palencia, Palencia
  - Vigo, Pontevedra
  - Langreo, Principality of Asturias
  - Soria, Soria
  - Reus, Tarragona
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Bilbao, Vizcaya
  - Vitoria-Gasteiz, Vizcaya
- United Kingdom (15):
  - Belfast
  - Bristol
  - Cambridge
  - Cheshire
  - Cornwall
  - Coventry
  - Essex
  - Glasgow
  - Hemel Hempstead
  - Lincolnshire
  - Norfolk
  - Nottingham
  - Stoke-on-Trent
  - Walsall
  - Wolverhampton

REFERENCES:
- [Derived] Domenech C, Pastore A, Altamura AC, Bernasconi C, Corral R, Elkis H, Evans J, Malla A, Margari F, Krebs MO, Nordstroem AL, Zink M, Haro JM. Correlation of Health-Related Quality of Life in Clinically Stable Outpatients with Schizophrenia. Neuropsychiatr Dis Treat. 2019 Dec 20;15:3475-3486. doi: 10.2147/NDT.S218578. eCollection 2019. PMID 31908462
- [Derived] Franklin M, Mukuria C, Mulhern B, Tran I, Brazier J, Watson S. Measuring the Burden of Schizophrenia Using Clinician and Patient-Reported Measures: An Exploratory Analysis of Construct Validity. Patient. 2019 Aug;12(4):405-417. doi: 10.1007/s40271-019-00358-x. PMID 30820841
- [Derived] Domenech C, Bernasconi C, Moneta MV, Nordstroem AL, Cristobal-Narvaez P, Vorstenbosch E, Cobo J, Ochoa S, Haro JM. Health-related quality of life associated with different symptoms in women and in men who suffer from schizophrenia. Arch Womens Ment Health. 2019 Jun;22(3):357-365. doi: 10.1007/s00737-018-0896-0. Epub 2018 Aug 7. PMID 30088146